CLINICAL TRIAL: NCT00579605
Title: Motivational Interviewing to Promote Sustained Breastfeeding (Native American Women)
Brief Title: Motivational Interviewing to Promote Sustained Breastfeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0273-06-FB; UNMC MIHERO Internal Grant (Other Grant/Funding Number: University of Nebraska Medical Center)
Record Dates: First submitted 2007-12-19; First posted 2007-12-24 (Estimated); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Breastfeeding
Keywords: Breastfeeding; Self-efficacy; Motivational Interviewing
MeSH Terms: conditions — Breast Feeding | interventions — Motivational Interviewing; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 Motivational Interviewing (Experimental): 1 intervention group 1 attention intervention group Behavioral: Motivational Interviewing Client-centered strategy that may decrease ambivalence in behavior performance
  Interventions: Behavioral: Motivational Interviewing

INTERVENTIONS:
Behavioral: Motivational Interviewing — Client-centered strategy that may decrease ambivalence in behavior performance with attention intervention (infant safety) on: a) breastfeeding self-efficacy, b) intended length of breastfeeding, and c) duration of breastfeeding.
  Other Names: Counseling

SUMMARY:
1. Evaluate the cultural appropriateness of an intervention protocol related to: a) motivational interviewing technique; b) stool, urine, and breast milk sample collection; and c) infant breastfeeding test weight procedure.
2. Compare Motivational Interviewing with an attention intervention (infant safety) on: a) breastfeeding self-efficacy, b) intended length of breastfeeding, and c) duration of breastfeeding.
3. Examine urine samples of infants for the presence of the inflammatory cytokine (LTE4) and evaluate fecal and breast milk samples of infants for human milk oligosaccharide levels.

DETAILED DESCRIPTION:
The incidence of asthma, the most common serious chronic inflammatory disease among children, is rising each year. Therefore nursing interventions aimed at promoting infant immunity and mitigating factors to which the infant may be exposed may reduce the complications of this chronic illness. Breastfeeding is an ideal initial prevention strategy that strengthens the infant's immune system. In addition, the identification of biomarkers that reflect infant immune response sets the stage for the evaluation of nursing interventions targeted to decrease the impact of this chronic inflammatory disease. Although more mothers currently initiate breastfeeding, they do not sustain breastfeeding for the recommended 6 to 12 months. In general, Native American mothers' breastfeed for a shorter period of time and mothers in rural setting have fewer resources to support breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for mothers include ≥ 19 years of age and enrolled in Northern Plains Healthy Start program.
* Inclusion criteria for infants are birth weight of > 2500 gms, > 37 weeks gestation, a bilirubin of 15 mg%, and no NICU admission to provide a sample of stable infants.

Exclusion Criteria:

* Mothers who report that they will not breastfeed will be excluded.
* Infants with a birth weight < 2500 gms, are < 37 weeks gestation, or diagnosed with any significant health problems, significant postnatal problems requiring NICU admission, symptoms of drug withdrawal, or a bilirubin > 15 mg% will be not be recruited for the study.

Ages: 17 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2006-09-06 (Actual); Study Completion 2007-12-01 (Actual)

PRIMARY OUTCOMES:
Days of any breastfeeding | From delivery to 6 months after birth
  Number of days of any breastfeeding

SECONDARY OUTCOMES:
Increased Breastfeeding self-efficacy | From birth to 6 months after delivery
  Self-reported maternal satisfaction with breastfeeding
Increased intention to breastfeed for 6 months | From birth to 6 months
  Self-reported maternal intention to breastfeed for a 6 month period

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Wilhelm, RNC, PhD, Principal Investigator — University of Nebraska Medical Center, College of Nursing